CLINICAL TRIAL: NCT04756947
Title: Epidemiological Study of Pediatric Pelvic Injuries
Brief Title: Pediatric Pelvic Injuries - Epidemiology and Demography
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government); University Hospital Pilsen (Other)
Responsible Party: Principal Investigator, Valer Dzupa, Clinical Professor, Charles University, Czech Republic
Other Study IDs: Pediatric Pelvis 01
Record Dates: First submitted 2021-02-09; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Pelvis Injury; Child, Only

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pelvic injury: Paediatric patients (age ≤ 18 years) with a single pelvic bone fracture or pelvic ring injury, excluding pathological fractures.
  Interventions: Procedure: surgical treatment according to standard indication criteria; Procedure: conservative treatment according to standard indication criteria
- Pelvic and acetabular injury: Paediatric patients (age ≤ 18 years) with a combined pelvic and acetabular injury or an isolated acetabular fracture, excluding pathological fractures.
  Interventions: Procedure: surgical treatment according to standard indication criteria; Procedure: conservative treatment according to standard indication criteria

INTERVENTIONS:
Procedure: surgical treatment according to standard indication criteria — internal fixation according to standard indication criteria
Procedure: conservative treatment according to standard indication criteria — conservative therapy according to standard indication criteria

SUMMARY:
A retrospective epidemiological study of pediatric pelvic injury from level 1 trauma centre.

Hypothesis: In the pediatric population, majority of pelvic injuries is of type A according to AO/OTA (Arbeitsgemeinschaft für Osteosynthesefragen/Orthopaedic Trauma Association) classification, the treatment is mostly conservative and complications of injury and treatment are less common than in adults.

DETAILED DESCRIPTION:
Study design: Retrospective analysis (13 years), excluding pathological fractures. AO/OTA type, epidemiological data, mode of treatment, and complications were recorded. Data were analyzed using the Fisher exact test and the Wilcoxon test.

ELIGIBILITY:
Inclusion Criteria of primary study group:

* Age ≤ 18 years
* Single pelvic bone fractures or pelvic ring injuries

Inclusion Criteria of secondary study group:

* Age ≤ 18 years
* Combined pelvic and acetabular injuries
* Isolated fractures of the acetabulum

Exclusion Criteria:

* Pathological fractures

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 358 patients (243 boys, 115 girls), mean age (SD) 14.1 ± 3.0 years
Sampling Method: Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Epidemiological study of pediatric pelvic trauma | Follow-up of each patient for minimum 12 months.
  1. The overall incidence of pelvic ring injury per 100,000 children per year.
  2. The overall incidence of isolated acetabular fractures per 100,000 children per year.
  3. The overall incidence of combined pelvic ring and acetabular injuries per 100,000 children per year.

SECONDARY OUTCOMES:
Demographical study of pediatric pelvic trauma | Follow-up of each patient for longer then 12 months.
  1. Comparison of the incidence of observed injuries by sex.
  2. Comparison of the incidence of observed injuries according to the severity of trauma (single trauma vs. multiple trauma).
  3. The incidence of the types of pelvic ring injury (according to AO/OTA classification) per 100,000 children per year.

CONTACTS AND LOCATIONS:
Overall Officials: Valer Dzupa, MD, Study Chair — Charles University, Czech Republic

IPD SHARING:
Plan to Share IPD: No
Patients´ personal data will not be shared. The study results will be shared when published in a medical journal.

REFERENCES:
- [Background] DeFrancesco CJ, Sankar WN. Traumatic pelvic fractures in children and adolescents. Semin Pediatr Surg. 2017 Feb;26(1):27-35. doi: 10.1053/j.sempedsurg.2017.01.006. Epub 2017 Jan 5. PMID 28302282
- [Background] Tosounidis TH, Sheikh H, Giannoudis PV. Pelvic Fractures in Paediatric Polytrauma Patients: Classification, Concomitant Injuries and Early Mortality. Open Orthop J. 2015 Jul 31;9:303-12. doi: 10.2174/1874325001509010303. eCollection 2015. PMID 26312114